CLINICAL TRIAL: NCT00888719
Title: A Prospective, Randomized, Double Blinded, Multicenter and Therapeutic Exploratory Study to Comparatively Assess Efficacy and Safety of CWP-0403 in Type 2 Diabetes Patients Who Are Insufficiently Controlled by Diet and Exercise.
Brief Title: Therapeutic Exploratory Study of CWP-0403
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Hyung kyu, Park, ChoongWae Pharma Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CWP-SKD-201
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CWP-0403 50mg (Experimental)
  Interventions: Drug: CWP-0403 50mg
- CWP-0403 100mg (Experimental)
  Interventions: Drug: CWP-0403 100mg
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CWP-0403 100mg — 100mg/tablet, Twice a day, 1 tablet at a time for 12 weeks
  Arms: CWP-0403 100mg
Drug: placebo — Tablet not containing CWP-0403 and indistinguishable from CWP-0403 50mg, 100mg tablets.
  Twice a day, 1 tablet at a time for 12 weeks
  Arms: placebo
Drug: CWP-0403 50mg — 50mg/tablet, Twice a day, 1 tablet at a time for 12 weeks
  Arms: CWP-0403 50mg

SUMMARY:
Objective of the trial is to assess dose-dependency, efficacy and safety and to estimate optimum dosage for confirmatory study of CWP-0403 50mg, 100mg given twice daily for 12 weeks to type 2 diabetes patients who are insufficiently controlled by diet and exercise in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age of≥25 and <75 with typeⅡ DM patients
* Patients whose level of HbA1c is over 7.0% and less than 10% within 4weeks of screening registration
* In spite of dietary and exercise treatment over 8weeks, the level of HbA1c is over 6.5% and less than 10%.
* BMI between 20kg/㎡ and 40kg/㎡
* Out patients
* patients who agree the trial participation with written informed consent

Exclusion Criteria:

* TypeⅠDM, Gestational diabetes.
* Patients who are being treated with insulin
* Fasting glucose level over 250mg/dL
* Patients who are not compliant with dietary and exercise treatment during 8 weeks of screening period. (Evaluated "Bad" and worse)
* Severe hepatic dysfunctions (i.e.: uncompensated hepatic cirrhosis)or AST or ALT level over 2.5times as high as UNL on screening visit.
* Severe renal dysfunctions (i.e.: renal failure) or serum creatinine level over 1.5mg/dl
* Severe cardiac dysfunction(i.e.: heart failure ) or history of myocardial infarction within 6months of screening
* Chronic pulmonary disease or pulmonary infarction
* Pancreatitis patients
* Patients who are being treated for life threatening disease such as cancer, severe trauma or infection.
* Uncontrollable diabetic complications(neuropathy, retinopathy, nephrosis)
* Severe ketosis or experience of diabetic coma
* Intestinal disease affecting digestion or absorption or history of GI dissection surgery except for appendectomy.
* Pregnant, expecting to be pregnant or nursing female
* Excessive alcohol consumption (Over 80g of alcohol/day: Over 1 bottle of 360ml Soju/day)
* Participants of other clinical trials within 3 months of screening
* Patients medicated with following non-concomitant medications Insulins or oral antidiabetics Oral (for more than 1 week) or IV corticosteroids (External and inhaled corticosteroids excluded) appetite suppressant exenatide or other GLP-1 analogues Other medications in development
* Hypersensitive or intolerance to DPP4 inhibitory
* patients who are decided to be inappropriate for this trial subject by the investigators

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c before and after treatment | 12 weeks

SECONDARY OUTCOMES:
HbA1c target achievement rate(Ratio of the patients with HbA1c lower than 6.5% or 7%) | 12 weeks
Fasting blood glucose level change and rate of change | 12 weeks
Serum insulin, serum C-peptide level change | 12 weeks
HOMA-R and HOMA-β change rate | 12 weeks
Triglyceride, LDL-cholesterol and HDL-cholesterol change | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: KunHo Yoon, Principal Investigator — The Catholic University of Korea
Locations (10):
- South Korea (10):
  - Chonbuk National University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Gachon Medical School Gil Medical Center, Seoul
  - Inha University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyungpook National University Hospital, Seoul
  - Seoul National University Bundang Hopital, Seoul
  - The Catholic University of Korea, Holly Family Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Seoul